CLINICAL TRIAL: NCT06049043
Title: Testing Preliminary Effectiveness of a Community Health Worker (CHW) Training Program to Support African American and Latino Male Caregivers of Older Adults
Brief Title: Testing Preliminary Effectiveness of a Community Health Worker (CHW) Training Program on Caregiving
Acronym: IN-HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KDH Research & Communication (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-02-10
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Caregiver Burnout
Keywords: Male; Black or African American; Hispanic or Latino; Feasibility Studies
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention to Help Orient Men to Excel (IN-HOME) (Experimental): Professional development training for CHWs on African American and Latino male caregiver needs
  Interventions: Other: Intervention to Help Orient Men to Excel (IN-HOME)
- Control (Other): AARP's English "Care at Home" resource webpage
  Interventions: Other: AARP's English "Care at Home" resource webpage

INTERVENTIONS:
Other: Intervention to Help Orient Men to Excel (IN-HOME) — A multi module online training
  Arms: Intervention to Help Orient Men to Excel (IN-HOME)
Other: AARP's English "Care at Home" resource webpage — Caregiver information from the American Association of Retired Persons
  Arms: Control

SUMMARY:
Two arm study, experimental and control, to explore the impact of an online training program to prepare community health workers (CHWs) conduct effective outreach to support African American and Latino male caregivers of older adults.

DETAILED DESCRIPTION:
The investigators used a randomized, two-group, pretest/posttest design to test the efficacy of the IN-HOME prototype and explore the following research question: To what extent did exposure to the IN-HOME prototype relate to positive changes in Community Health Workers' (CHWs') knowledge, skills, and perceived self-efficacy to conduct outreach to African American and Latino male caregivers of older adults?

The community-focused and community-based approach of the intervention included an evaluation that required strategies to address gender preferences for resources and providing care and cultural awareness to understand the communities of focus. The evaluation recognized additional barriers such as racial/ethnic group historical experiences and racism that effects the groups health outcomes and health care interactions. To ensure that the approach was culturally appropriate and the materials were culturally relevant, the investigators worked with caregiver and health disparities researchers and CHW practitioners to create an advisory committee of experts that provided input into the development of the intervention to empower CHWs to conduct outreach to African American and Latino male caregivers. The PI, with input from the advisory committee, developed necessary research materials, including the recruitment protocols, evaluation instrumentation, and human subjects consent materials. The PI also outlined the appropriate statistical analysis methods. All procedure documents were reviewed by the Institutional Review Board before the evaluation launch.

The investigators recruited participants through evaluation partners who disseminated the study information to CHWs via electronic notifications and flyers. Evaluation partners included sites with CHW-related programs and CHW organizations such as, the Virginia CHW Association, the Dallas-Fort Worth CHW Organization, Connection Health, and the Hispanic Health Initiative Incorporated. The notification provided information about the goal of the study, participant eligibility, and a link to an interest and eligibility form. After a potential participant completed the interest and eligibility form and determined as eligible for the project, they received a link to a consent form that was located on a secure online platform.

CHWs were randomly assigned to the intervention or control group after consent and enrollment in the study. All participants completed an online pretest survey. The intervention group was exposed to IN-HOME and completed an online posttest survey two weeks after completing the IN-HOME modules. The control group participants were not exposed to the IN-HOME program but were asked to review the AARP's English "Care at Home" resource webpage. The control group participants completed a posttest two weeks after completing the pretest. Participant responses to pretest and posttest survey measures were linked using non-personal identifiers.

The investigators downloaded and exported the data from the online data collection system into an encrypted Excel file and imported the raw data into STATA. The investigators matched the pretest and posttest responses using the random assigned identifiers and conduct analyses to test for the effect of IN-HOME exposure on changes in CHWs' knowledge, skills, and self-efficacy to conduct outreach to African American and Latino male caregivers. Effectiveness measure for intervention feasibility was statistically significant differences between pretest and posttest for knowledge and self-efficacy measures among the intervention group participants.

ELIGIBILITY:
Inclusion Criteria:

* Must self-identify as working as a community health worker
* Must be actively employed conducting community-based outreach at an organization (paid or volunteer)
* Must be 18 years of age or older
* Must live in the United States

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Twombly, PhD, Study Chair — KDH Research & Communication
Locations (1):
- KDH Research & Communication, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Started | 55 | 52
Completed | 44 | 43
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 42 | 83
  >=65 years | 3 | 1 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 10 | 13 | 23
  Sex: Female | 34 | 29 | 63
  Sex: Prefer not answer | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 31 | 65
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Education level [Count of Participants; unit: Participants]
  High school diploma/GED | 6 | 4 | 10
  Some college | 7 | 8 | 15
  College degree | 20 | 17 | 37
  Master's degree | 10 | 13 | 23
  Professional degree | 1 | 1 | 2
Years of CHW experience [Count of Participants; unit: Participants]
  6 to 11 months | 4 | 6 | 10
  1 to 2 years | 18 | 13 | 31
  3 to 4 years | 3 | 11 | 14
  5 or more years | 17 | 13 | 30
  Prefer not to answer | 2 | 0 | 2
Type of CHW [Count of Participants; unit: Participants]
  Paid | 25 | 24 | 49
  Volunteer | 7 | 5 | 12
  Both | 8 | 13 | 21
  Prefer not answer | 4 | 1 | 5
Hours training [Count of Participants; unit: Participants]
  None | 2 | 0 | 2
  1 to 5 hours | 3 | 3 | 6
  6 to 10 hours | 7 | 5 | 12
  11 to 15 hours | 0 | 5 | 5
  16+ hours | 32 | 30 | 62
Trained in caregiving for older adults [Count of Participants; unit: Participants] — Have you previously received training about caregiving for older adults?
  Participants
    Yes | 25 | 19 | 44
    No | 18 | 21 | 39
    I don't know | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Pretest
Description: We asked participants 16 identically worded knowledge-based multiple-choice questions during the pretest and posttest. For each participant, we averaged their correct scores from these knowledge questions, resulting in a score that ranged from 0 to 100, with 0 as the minimum score and 100 as the maximum score. Higher scores indicate better outcomes. We then averaged these individual scores across all participants to create a composite average knowledge score for group comparisons, also ranging from 0 to 100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 40 | 39
score on a scale | 79.84 (23.02) | 84.94 (16.14)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = -5.09, 95% CI 2-sided [-14.02 to 3.84], Standard Error of Mean 0.04

2. Primary Outcome: Skills Pretest
Description: We asked participants eight identically worded skills-based multiple-choice questions at pretest and posttest. For each participant, we averaged their correct scores from these skills questions, resulting in a score that ranged from 0 to 100, with 0 as the minimum score and 100 as the maximum score. Higher scores indicate better outcomes. We then averaged these individual scores across all participants to create a composite average skills score for group comparisons, also ranging from 0 to 100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 42 | 41
score on a scale | 80.36 (23.29) | 84.15 (20.73)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-13.43 to 5.85], Standard Error of Mean 4.84

3. Primary Outcome: Self-efficacy Pretest
Description: We asked participants 15 identically worded questions relating to their perceived self-efficacy/confidence in providing outreach to male caregivers. Each answer choice was a 10-point confidence rating scale, ranging from 1 (not very confident) to 10 (very confident), with higher scores indicating better outcomes. We averaged self-efficacy scores across all self-efficacy questions for each participant, then averaged these scores across all participants for group comparisons.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 38 | 41
score on a scale | 7.25 (2.00) | 7.03 (1.93)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.62, t-test, 2 sided; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.66 to 1.10], Standard Error of Mean 0.44

4. Primary Outcome: Knowledge Posttest
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 43 | 42
score on a scale | 89.83 (20.37) | 83.48 (20.61)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = 6.34, 95% CI 2-sided [-2.50 to 15.18], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.28, Regression, Linear; Controlled for participant characteristics at baseline; Slope = -0.05, 95% CI 2-sided [-0.13 to 0.04], Standard Error of Mean 0.04

5. Primary Outcome: Skills Posttest
Description: as for outcome 2
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 44 | 42
score on a scale | 83.24 (21.89) | 81.25 (21.43)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.67, t-test, 2 sided; Mean Difference (Final Values) = 1.98, 95% CI 2-sided [-7.31 to 11.28], Standard Error of Mean 4.67
Statistical Analysis 2: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.69, Regression, Linear; Controlled for participant characteristics at baseline; Slope = -0.02, 95% CI 2-sided [-0.12 to 0.08], Standard Error of Mean 0.05

6. Primary Outcome: Self-efficacy Posttest
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 40 | 40
score on a scale | 8.55 (1.17) | 8.01 (1.63)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.09 to 1.18], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.71, Regression, Linear; Controlled for participant characteristics at baseline; Slope = -0.13, 95% CI 2-sided [-0.86 to 0.59], Standard Error of Mean 0.36

7. Primary Outcome: Preparedness Posttest
Description: We asked participants six identically worded questions relating to their perceived preparedness to deliver male caregiver outreach at pretest and posttest. Each answer choice was a 10-point confidence rating scale, ranging from 1 (not at all prepared) to 10 (very much prepared), with higher scores indicating better outcomes. We averaged scores from each preparedness question for each participant, then averaged these scores across all participants for group comparisons.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 41 | 41
score on a scale | 8.61 (1.28) | 8.02 (1.74)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-0.07 to 1.27], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.39, Regression, Linear; Controlled for participant characteristics at baseline; Slope = -0.36, 95% CI 2-sided [-1.21 to 0.48], Standard Error of Mean 0.42

8. Secondary Outcome: Satisfaction Composite Scores at Posttest
Description: We asked intervention group participants five questions about their satisfaction with IN-HOME at posttest. All five satisfaction questions were ratings assessing the participants' perceptions of ease, relevance, engagement, usefulness, and likeliness to tell others about IN-HOME. Each answer choice ranged from 1 to 10, with 10 representing the highest and 1 representing the lowest rating. We averaged satisfaction ratings across all five questions for each intervention participant and averaged these scores across all intervention participants to create a single composite score ranging from 1 to 10, with higher scores indicating higher satisfaction.
Time Frame: 2/3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME)
Number analyzed (Participants) | 43
score on a scale | 8.91 (1.33)

9. Primary Outcome: Preparedness Pretest
Description: as for outcome 7
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
Number analyzed (Participants) | 41 | 42
score on a scale | 7.05 (1.98) | 7.12 (2.07)
Statistical Analysis 1: Comparison: Intervention to Help Orient Men to Excel (IN-HOME) vs Control; Test type: Superiority; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.95 to 0.82], Standard Error of Mean 0.22

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Intervention to Help Orient Men to Excel (IN-HOME) | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT06049043/Prot_SAP_000.pdf